CLINICAL TRIAL: NCT04361721
Title: Neurophysiological, Biomolecular and Psychological Aspects of Erenumab Treatment in Chronic Migraine: an Open Label, Hypothesis Generator Study
Brief Title: Neurophysiological, Biomolecular and Psychological Aspects of Erenumab Treatment in Chronic Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EreCM2019
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2020-04

CONDITIONS: Chronic Migraine
Keywords: Spinal sensitization; Biomarkers; Anti CGRP monoclonal antibodies; Migraine phenotypes
MeSH Terms: interventions — erenumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA concentration was determined by absorbance at 230 and 280 nm using the NanoDrop Spectrophotometer (Euroclone Milano). Synthesis of cDNA was performed by using MirXMirna First strand Synthesis (Takara-Diatech, Jesi-An Italy) and TB Green q-Rt PCR is used (Takara-Diatech, Jesi-An Italy) to determine expression levels of miRNA-34a-5p and miRNA-382-5p. The denaturation was performed at 95°C and the amplification was performed through two-step cycling (95-60°C) for 40 cycles with a Light Cycler 480 Instrument RT-PCR Detection System (Roche, Milan, Italy). Target gene expression levels was normalized with U6 (a type of small nuclear RNA), used as housekeeping gene. Gene expression levels were calculated according to 2-∆Ct = 2 - (Ct gene - Ct housekeeping gene) formula by using Ct values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Chronic migraine patients: Three monthly administration of erenumab 70 mg subcutaneously.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — First injection of erenumab 70 mg subcutaneously was administered in hospital. The second injection of erenumab 70 mg was administered in hospital after 28 days, while the third and last dose of erenumab 70 mg was self-administered at home by the patients themselves after an additional 28-day interval.

SUMMARY:
Monoclonal antibodies (mABs) targeting calcitonin gene-related peptide (CGRP) proved effective in the preventive treatment of episodic and chronic migraine as well as in difficult-to-treat patients such as those who had previously failed multiple prevention treatments or those with associated medication overuse (MO).

A characteristic dysfunction in Chronic Migraine (CM) is sensitization, occurring peripherally in the trigeminovascular system but then spreading to the central nervous system, where it manifests with an increased neuronal excitability in multiple areas. Several neurophysiological studies in CM patients have demonstrated the occurrence of central sensitization in the brain as well as at the spinal level.

MicroRNAs (miRNAs) are involved in the generation and maintenance of chronic pain. Current evidence suggests that specific miRNAs may also play a role in migraine, thus representing possible biomarkers of the disease. A previous study reported an upregulation of miR-34a-5p and miR-382-5p, implicated in the regulation of GABAergic signaling and IL-10 gene expression respectively, during migraine attacks.

The aim of this open label, hypothesis generating study is the evaluation of the impact of erenumab treatment on neurophysiological, biomolecular and psychological aspects in a representative cohort of CM patients who had previously failed at least 2 preventive treatments.

DETAILED DESCRIPTION:
This study consisted of a first screening visit with a Neurologist of the Headache Science Centre of the IRCCS Mondino Foundation, during which a full neurological and general examination was performed, and the data collected on the routine headache diary used by all patients attending Mondino Foundation was checked to confirm inclusion/exclusion criteria.

If a patient fulfilled criteria, he/she was enrolled in a baseline observation period for a month. At the end of the baseline observation period (T0), if inclusion/exclusion criteria were still satisfied, patients completed the following procedures: recording of clinical and demographical features, vital signs evaluation, neurophysiological assessment and psycological interview based on DSM (The Diagnostic and Statical Manual of Mental Disorders), venous blood sampling, and compilation of a set of self-administered questionnaires about psychological state, health status and quality of life.

At T0, the patients were treated with the first dose of erenumab 70 mg subcutaneously.

After 28 days (4 full weeks), patients returned for the second visit (T1) to report clinical variables and adverse events. During T1, the second injection of erenumab 70 mg was administered, while a third and last dose of erenumab 70 mg was self-administered at home by the patients themselves after an additional 28-day interval (T2). The last visit of the study (T3) was then planned 56 days from T1, that was 28 days after the last dose of erenumab. At T3, the patients were tested with the same multi-disciplinary evaluation performed at T0: recording of clinical and demographical features, vital signs evaluation, neurophysiological assessment, venous blood sampling, and compilation of questionnaires concerning patients' psychological state, health status and quality of life.

Nociceptive withdrawal reflex measurements. The nociceptive withdrawal reflex (NWR) is considered an objective and solid neurophysiological technique for the study of spinal nociceptive transmission. The reflex was recorded in the lower limb according to a well validated procedure, in a quiet environment by an expert technician between 09:00 AM and 11:00 AM. Patients were in a comfortable position with their ankle flexed at 90° and knee flexed at 130°. The sural nerve was stimulated electrically behind the lateral malleolus with a pair of Ag/AgCl surface electrodes. The electrical stimulation was made of 5 consecutive squared pulses (1 ms, 200 Hz), randomly delivered every 60-120 seconds. The electromyographic sweep (Synergy, Medelec, United Kingdom) was recorded from the capitis brevis of the homolateral biceps femoris with a pair of Ag/AgCl surface electrodes. A staircase method was used for all the threshold evaluations, and the intensity was increased by 0.3 mA per step. The recording parameters were: analysis time 300 ms, sensitivity 20 mV, and filter bandpass 3 to 3000 Hz.

The investigators first evaluated the single stimulus reflex threshold of the NWR (RTh), defined as the lowest intensity (mA) able to induce 3 consecutive stable muscular responses of at least 20 mV and 10 ms. They also evaluated the average AUC (Area Under the Curve - mV x ms), the average latency (ms), and the subjective pain perception rated on a 0-10 points visual analogue scale (VAS-RTh).

Then the investigators evaluated the temporal summation threshold (TST), by means of a train of 5 electrical stimuli at a frequency of 2 Hz. TST was defined as the lowest intensity (mA) able to elicit 3 consecutive stable muscular responses of at least 20 mV and 10 ms in the fourth and fifth electromyographic sweeps. They also evaluated the subjective pain perception of the first (VAS-TST-1) and fifth (VAS-TST-5) stimulus of the TST on a 0-10 points visual analogue scale.

MicroRNAs expression. The microRNA expression was evaluated by real-time reverse transcription (RT) PCR in peripheral blood mononuclear cell (PBMCs).

PBMCs isolation: blood samples (10 ml) was collected within ethylenediamine tetra-acetic acid containing tube from participants. The blood samples were diluted in 1:1 ratio with phosphate buffer saline (PBS) (Sigma). Diluted blood samples were slowly loaded into Ficoll separating solution (10 ml) (Sigma) and centrifuged at 800 g for 30 min at room temperature. PBMCs accumulated as the middle white monolayer, were washed twice in sterile PBS at 300 g for 15 min. After washing, PBMCs were pelleted and stored at -80° C until use.

MicroRNAs gene expression: isolation of RNA from PBMCs was carried out using the Direct-zol RNA Mini prep plus (Zymo Research). RNA concentration was determined by absorbance at 230 and 280 nm using the NanoDrop Spectrophotometer (Nanodrop™ Thermo Fisher Scientific, Euroclone Milano). Synthesis of cDNA was performed by using MirXMirna First strand Synthesis (Takara-Diatech, Jesi-An Italy) and TB Green q-Rt PCR is used (Takara-Diatech, Jesi-An Italy) to determine expression levels of miRNA-34a-5p and miRNA-382-5p. The denaturation was performed at 95°C and the amplification was performed through two-step cycling (95-60°C) for 40 cycles with a Light Cycler 480 Instrument RT-PCR Detection System (Roche, Milan, Italy). Target gene expression levels was normalized with U6 (a type of small nuclear RNA), used as housekeeping gene. Gene expression levels were calculated according to 2-∆Ct = 2 - (Ct gene - Ct housekeeping gene) formula by using Ct values.

Disability and psychological evaluations.

The battery included evaluations for:

4) Migraine-related disability and associated features:

* the Migraine Disability Assessment (MIDAS) test: 0-5 (grade I): minimal disability, 6-10 (grade II): mild disability, 11-20 (grade III): moderate disability, 21-40 (grade IVa): severe disability, 41 and higher (grade IVb): very severe disability;
* the Headache Impact Test-6 (HIT-6): 49 or less: no impact, 50-55: some impact, 56-59: substantial impact, 60-78 severe impact;
* Nociceptive Rating Scale for the assessment of average intensity of migraine pain: 0 no pain - 10 very severe;
* Allodynia Symptom Checklist (ASC-12): 0-3: mild cutaneous allodynia, 6-8: moderate cutaneous allodynia, 9 and higher: severe cutaneous allodynia.

  5) Quality of life:
* the Migraine-Specific Quality-of-Life Questionnaire (MSQ): 14-item assessment, with each item rated on a 6-point scale (ranging from "none of the time" to "all of the time"). Raw scores are then transformed to a 100-point scale, with higher scores indicating better quality of life;
* Short Form Health Survey (SF-36): 11-item assessment referring to two main sub-domains, namely the Mental Component Summary (MCS), and the Physical Component Summary (PCS);
* HEALTH 0-100: patients were asked to score on a scale range of 0-100 their general health status at the precise moment of evaluation.

  6) Psychological State:
* Hospital Anxiety and Depression Scale (HADS): a 14-items questionnaire on a 4-point (0-3) Likert scale assessing symptoms of anxiety and depression. A score of 8 or higher in the two different domains is considered significant for anxiety and/or depression;
* Leeds Dependence Questionnaire (LDQ): a 10-item instrument on 0-3 scale to measure dependence upon a variety of substances. No cut-off score indicative of dependence has been established;
* Toronto Alexithymia Scale (TAS-20): a 20-item questionnaire on a 5-point (1-5) Likert scale assessing alexithymia traits, i.e., individuals' difficulty in expressing their own feelings in words. A score of 61 or higher was considered significant for the presence of alexithymia;
* Childhood trauma questionnaire: including 13 items referring to different types of childhood traumas that were considered in term of total number of traumatic experiences;
* Stressful life-events questionnaire: consisting in a list of 58 stressful life events (e.g., moving, divorce, new work, dismissal, etc.). Patients were requested to tick those events that had occurred to them in the last 10 years.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65 years
* history of CM or CM+MO for at least 12 months prior to enrollment [10]
* previous failure of at least two different pharmacological classes of preventive therapies

Exclusion Criteria:

* other neurologic or neuropsychiatric diseases
* other chronic painful syndromes
* other types of primary or secondary headaches
* use of more than one preventive medication at baseline
* previous reported adverse reaction to latex
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty patients, affected by CM or CM+MO according to the International Classification of Headache Disorders (ICHD) -3 criteria were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Spinal sensitization | Change in TST (mA) at T3 (12 weeks later) when compared to baseline (T0)
  Measured by the temporal summation threshold (TST) of the nociceptive withdrawal reflex

SECONDARY OUTCOMES:
Spinal sensitization | Change in RTh (mA) at T3 (12 weeks later) when compared to baseline (T0)
  Measured by the single stimulus reflex threshold (RTh) of the nociceptive withdrawal reflex.
Inflammatory biomarker profile | Change in miR-382-5p at T3 (12 weeks later) when compared to baseline (T0)
  Measured by plasma levels of miR-382-5p
inflammatory biomarker profile | Change in miR-34a-5p at T3 (12 weeks later) when compared to baseline (T0)
  Measured by plasma levels of miR-34a-5p
Migraine Disability Assessment (MIDAS) | Change in MIDAS score at T3 (12 weeks later) when compared to baseline (T0)
  Migraine-related disability as measured by MIDAS test: 0-5 (grade I): minimal disability, 6-10 (grade II): mild disability, 11-20 (grade III): moderate disability, 21-40 (grade IVa): severe disability, 41 and higher (grade IVb): very severe disability.
Headache Impact Test-6 (HIT-6) | Change in HIT-6 score at T3 (12 weeks later) when compared to baseline (T0)
  Migraine-related disability as measured by HIT-6 test: 49 or less: no impact, 50-55: some impact, 56-59: substantial impact, 60-78 severe impact.
Allodynia Symptom Checklist (ASC-12) | Change in ASC-12 score at T3 (12 weeks later) when compared to baseline (T0)
  Migraine-related disability as measured by ASC-12 test: 0-2: none; 3-5: mild; 6-8: moderate; 9 or more: severe.
Migraine-Specific Quality-of-Life Questionnaire (MSQ) | Change in MSQ2 score at T3 (12 weeks later) when compared to baseline (T0)
  Quality of life measured by MSQ. 14-item assessment, with each item rated on a 6-point scale (ranging from "none of the time" to "all of the time"). We evaluated 3 scores, namely Role Function-Restrictive (RR), Role Function- Preventive (RP), and Emotional Function (EF). Raw scores have been transformed to a 100-point scale, with higher scores indicating better quality of life.
Short Form Health Survey (SF-36) | Change in SF-36 score at T3 (12 weeks later) when compared to baseline (T0)
  Quality of life measured by SF-36. 36-item assessment that gives us information about 8 different domains: physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items)
Hospital Anxiety and Depression Scale (HADS) | Change in HADS score at T3 (12 weeks later) when compared to baseline (T0)
  Psychological state as measured by HADS. a 14-items questionnaire on a 4-point (0-3) Likert scale assessing symptoms of anxiety and depression. A score of 8 or higher in the two different domains is considered significant for anxiety and/or depression;
Leeds Dependence Questionnaire (LDQ) | Change in LDQ score at T3 (12 weeks later) when compared to baseline (T0)
  Psychological state measured by LDQ. It is a self-completion 10-item instrument to measure dependence upon a variety of substances. No cut-off score indicative of dependence has been established
Toronto Alexithymia Scale (TAS-20) | Change in TAS-20 score at T3 (12 weeks later) when compared to baseline (T0)
  Psychological state measured by TAS-20. It is a 20-item questionnaire on a 5-point (1-5). Likert scale assessing alexithymia traits, i.e., individuals' difficulty in expressing their own feelings in words. A score of 61 or higher was considered significant for the presence of alexithymia.
Percentage of patients with positive clinical outcome | Percentage of 30% Responder patients at T3 (12 weeks after T0)
  Measured by percentage of patients with a reduction in migraine days of a least 30% (30% Responder).
Percentage of patients with positive clinical outcome | Percentage of 50% Responder patients at T3 (12 weeks after T0)
  Measured by percentage of patients with a reduction in migraine days of a least 50% (50% Responder).

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, Principal Investigator — IRCCS Mondino Foundation
Locations (1):
- IRCCS Mondino Foundation, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charles A, Pozo-Rosich P. Targeting calcitonin gene-related peptide: a new era in migraine therapy. Lancet. 2019 Nov 9;394(10210):1765-1774. doi: 10.1016/S0140-6736(19)32504-8. Epub 2019 Oct 23. PMID 31668411
- [Background] Ashina M, Tepper S, Brandes JL, Reuter U, Boudreau G, Dolezil D, Cheng S, Zhang F, Lenz R, Klatt J, Mikol DD. Efficacy and safety of erenumab (AMG334) in chronic migraine patients with prior preventive treatment failure: A subgroup analysis of a randomized, double-blind, placebo-controlled study. Cephalalgia. 2018 Sep;38(10):1611-1621. doi: 10.1177/0333102418788347. Epub 2018 Jul 8. PMID 29984601
- [Background] Tepper SJ, Diener HC, Ashina M, Brandes JL, Friedman DI, Reuter U, Cheng S, Nilsen J, Leonardi DK, Lenz RA, Mikol DD. Erenumab in chronic migraine with medication overuse: Subgroup analysis of a randomized trial. Neurology. 2019 May 14;92(20):e2309-e2320. doi: 10.1212/WNL.0000000000007497. Epub 2019 Apr 17. PMID 30996056
- [Background] Coppola G, Di Lorenzo C, Schoenen J, Pierelli F. Habituation and sensitization in primary headaches. J Headache Pain. 2013 Jul 30;14(1):65. doi: 10.1186/1129-2377-14-65. PMID 23899115
- [Background] De Icco R, Perrotta A, Grillo V, Cosentino G, Sances G, Sandrini G, Tassorelli C. Experimentally induced spinal nociceptive sensitization increases with migraine frequency: a single-blind controlled study. Pain. 2020 Feb;161(2):429-438. doi: 10.1097/j.pain.0000000000001726. PMID 31633594
- [Background] Andersen HH, Duroux M, Gazerani P. Serum MicroRNA Signatures in Migraineurs During Attacks and in Pain-Free Periods. Mol Neurobiol. 2016 Apr;53(3):1494-1500. doi: 10.1007/s12035-015-9106-5. Epub 2015 Feb 1. PMID 25636687
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Demartini C, Greco R, Zanaboni AM, Sances G, De Icco R, Borsook D, Tassorelli C. Nitroglycerin as a comparative experimental model of migraine pain: From animal to human and back. Prog Neurobiol. 2019 Jun;177:15-32. doi: 10.1016/j.pneurobio.2019.02.002. Epub 2019 Feb 13. PMID 30771365
- [Background] Sandrini G, Serrao M, Rossi P, Romaniello A, Cruccu G, Willer JC. The lower limb flexion reflex in humans. Prog Neurobiol. 2005 Dec;77(6):353-95. doi: 10.1016/j.pneurobio.2005.11.003. Epub 2005 Dec 28. PMID 16386347
- [Background] Schmittgen TD, Livak KJ. Analyzing real-time PCR data by the comparative C(T) method. Nat Protoc. 2008;3(6):1101-8. doi: 10.1038/nprot.2008.73. PMID 18546601
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Lipton RB, Bigal ME, Ashina S, Burstein R, Silberstein S, Reed ML, Serrano D, Stewart WF; American Migraine Prevalence Prevention Advisory Group. Cutaneous allodynia in the migraine population. Ann Neurol. 2008 Feb;63(2):148-58. doi: 10.1002/ana.21211. PMID 18059010
- [Background] Jhingran P, Osterhaus JT, Miller DW, Lee JT, Kirchdoerfer L. Development and validation of the Migraine-Specific Quality of Life Questionnaire. Headache. 1998 Apr;38(4):295-302. doi: 10.1046/j.1526-4610.1998.3804295.x. PMID 9595870
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Scalone L, Cortesi PA, Mantovani LG, Ciampichini R, Cesana G. Reference Eq-5d-3l and Eq-5d-5l Data From the Italian General Population. Value Health. 2014 Nov;17(7):A514-5. doi: 10.1016/j.jval.2014.08.1591. Epub 2014 Oct 26. No abstract available. PMID 27201592
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Raistrick D, Bradshaw J, Tober G, Weiner J, Allison J, Healey C. Development of the Leeds Dependence Questionnaire (LDQ): a questionnaire to measure alcohol and opiate dependence in the context of a treatment evaluation package. Addiction. 1994 May;89(5):563-72. doi: 10.1111/j.1360-0443.1994.tb03332.x. PMID 8044122
- [Background] Bagby RM, Parker JDA, Taylor GJ. Twenty-five years with the 20-item Toronto Alexithymia Scale. J Psychosom Res. 2020 Apr;131:109940. doi: 10.1016/j.jpsychores.2020.109940. Epub 2020 Jan 23. PMID 32007790
- [Background] Bottiroli S, Galli F, Viana M, Sances G, Tassorelli C. Traumatic Experiences, Stressful Events, and Alexithymia in Chronic Migraine With Medication Overuse. Front Psychol. 2018 May 14;9:704. doi: 10.3389/fpsyg.2018.00704. eCollection 2018. PMID 29867669
- [Derived] Bottiroli S, De Icco R, Vaghi G, Pazzi S, Guaschino E, Allena M, Ghiotto N, Martinelli D, Tassorelli C, Sances G. Psychological predictors of negative treatment outcome with Erenumab in chronic migraine: data from an open label long-term prospective study. J Headache Pain. 2021 Oct 2;22(1):114. doi: 10.1186/s10194-021-01333-4. PMID 34600468
- [Derived] De Icco R, Fiamingo G, Greco R, Bottiroli S, Demartini C, Zanaboni AM, Allena M, Guaschino E, Martinelli D, Putorti A, Grillo V, Sances G, Tassorelli C. Neurophysiological and biomolecular effects of erenumab in chronic migraine: An open label study. Cephalalgia. 2020 Oct;40(12):1336-1345. doi: 10.1177/0333102420942230. Epub 2020 Jul 26. PMID 32715736